CLINICAL TRIAL: NCT01495533
Title: Treatment of Coronary In-stent Restenosis by a Paclitaxel Coated AngioSculpt Scoring Balloon - a First-in-man Pilot Study
Brief Title: Paclitaxel-coated or Uncoated AngioSculpt Scoring Balloon Catheter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIM-DCA-01
Record Dates: First submitted 2011-12-13; First posted 2011-12-20 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: In-stent Arterial Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- uncoated AngioSculpt(R) (Active Comparator): Predilatation of coronary BMS-ISR with POBA followed by a AngioSculpt(R) scoring balloon (no drug coating)
  Interventions: Device: uncoated AngioSculpt(R)
- drug coated AngioSculpt(R) (Active Comparator): Predilatation of coronary BMS-ISR with POBA followed by a drug coated AngioSculpt(R) scoring balloon (paclitaxel 3.0 µg/mm²)
  Interventions: Combination Product: Drug coated AngioSculpt(R)

INTERVENTIONS:
Device: uncoated AngioSculpt(R) — Predilatation of coronary BMS-ISR with POBA followed by a AngioSculpt(R) scoring balloon (no drug coating)
  Arms: uncoated AngioSculpt(R)
Combination Product: Drug coated AngioSculpt(R) — Predilatation of coronary BMS-ISR with POBA followed by a drug coated AngioSculpt(R) scoring balloon (paclitaxel 3.0 µg/mm²)
  Arms: drug coated AngioSculpt(R)

SUMMARY:
The purpose of this study is to examine the treatment of coronary Bare Metal Stent restenosis with a drug coated AngioSculpt scoring balloon.

DETAILED DESCRIPTION:
Prospective, controlled, multicenter, randomized, single-blind trial. The aim is to examine the treatment of coronary Bare Metal Stent restenosis with a drug coated AngioSculpt scoring balloon. Patients are randomized to treatment by an AngioSculpt scoring balloon (no drug coating)or a drug coated AngioSculpt scoring balloon (paclitaxel 3.0 µg/mm²). Primary efficacy endpoint is late lumen loss in-segment at 6 months. Key secondary endpoints include procedural Success, MACE (cardiac death, target vessel myocardial infarction, and clinically driven target lesion revascularization at 6 months). Individual clinical endpoints include stent thrombosis (ARC), cardiac death, any death, target vessel myocardial infarction, any infarction, clinically driven target lesion revascularization, clinically driven target vessel revascularization, any revascularization.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* clinical evidence of stable or unstable angina or a positive functional study
* patients with ≤ 2 primary in-stent restenosis (ISR) lesions (≥ 70% diameter stenosis) within previously placed bare metal stents (BMS)

Exclusion Criteria:

* acute myocardial infarction within the past 72 hours
* chronic renal insufficiency with serum creatinine levels >2.0 mg per deciliter%
* known hypersensitivity or contraindications to aspirin, heparin, clopidogrel, ticlopidine or paclitaxel, and sensitivity to contrast media not amenable to premedication
* concomitant medical illness associated with a life-expectancy of less than two years
* stented segment length ≥30 mm, vessel diameter <2.5 mm, diameter stenosis <70%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
late lumen loss in-segment | 6 months
  angiographic late lumen loss in-segment assessed by quantitative coronary angiography

SECONDARY OUTCOMES:
Procedural Success | participants will be followed for the duration of hospital stay, an expected average of 2 days
  <50% final DS and the absence of in-hospital MACE
Major adverse cardiovascular events | 6 months
  the occurence of cardiac death, target vessel myocardial infarction, or clinically driven target lesion revascularization at 6 months (before planned control angiography)

CONTACTS AND LOCATIONS:
Locations (3):
- Danta Pazzanese Heart Institute, São Paulo, Brazil
- Germany (2):
  - Internal Medicine III, UKS, Homburg Saar
  - Herzzentrum Leipzig, Leipzig

REFERENCES:
- [Derived] Scheller B, Fontaine T, Mangner N, Hoffmann S, Bonaventura K, Clever YP, Chamie D, Costa R, Gershony G, Kelsch B, Kutschera M, Genereux P, Cremers B, Bohm M, Speck U, Abizaid A. A novel drug-coated scoring balloon for the treatment of coronary in-stent restenosis: Results from the multi-center randomized controlled PATENT-C first in human trial. Catheter Cardiovasc Interv. 2016 Jul;88(1):51-9. doi: 10.1002/ccd.26216. Epub 2015 Sep 2. PMID 26331782